CLINICAL TRIAL: NCT07191353
Title: Resistance Training and Rapamycin to Enhance Bone Formation in Postmenopausal Women
Acronym: StrongBone
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-520372-10-00
Record Dates: First submitted 2025-09-09; First posted 2025-09-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Osteopenia; Osteoporosis Risk
Keywords: Postmenopausal Women; Rapamycin; Bone formation; Muscle functions; Healthy aging
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Everolimus; Resistance Training

STUDY DESIGN:
Intervention Model Description: Phase 2, two-parallel, randomized, placebo-controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Treatment allocation to rapamycin or placebo is double-blinded, while allocation to training or no training will be known to participants and investigators, but masked to the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Everolimus (Experimental): Oral everolimus 5 mg once a week
  Interventions: Drug: Everolimus
- Everolimus and resistance training (Experimental): Oral everolimus 5 mg once a week plus resistance training RT 1 hour, 3 times weekly
  Interventions: Drug: Everolimus; Other: Resistance training
- Placebo (Placebo Comparator): Oral placebo once a week
  Interventions: Drug: Placebo
- Placebo and resistance training (Placebo Comparator): Oral placebo once a week plus resistance training RT 1 hour, 3 times weekly
  Interventions: Drug: Placebo; Other: Resistance training

INTERVENTIONS:
Drug: Everolimus — Everolimus 5 mg administered once weekly for 24 weeks
  Arms: Everolimus; Everolimus and resistance training
Drug: Placebo — Placebo administered once weekly for 24 weeks
  Arms: Placebo; Placebo and resistance training
Other: Resistance training — Resistance training 3 times a week for 24 weeks
  Arms: Everolimus and resistance training; Placebo and resistance training

SUMMARY:
The aim of the present clinical trial is to examine the effects of everolimus, resistance training, or their combination on bone and muscle health formation in elderly women aged 60-75 years. The main questions it aims to answer are:

Can rapamycin's analog (Everolimus), resistance training, or their combination, enhance bone formation and muscle functions in elderly women compared to non-treatment controls.

Participants will be randomized 1:1:1:1 to one of the following treatment regimens:

* Oral everolimus 5 mg once a week.
* Oral placebo once a week.
* Oral everolimus 5 mg once a week plus resistance training RT 1 hour, 3 times weekly.
* Oral placebo once a week plus resistance training RT 1 hour, 3 times weekly.

During the study there will be a total of 5-7 visits, where the participants will undergo the following:

* Blood samles
* DXA-, HRpQCT- (only Odense Universitetshospital) and MRI-scans
* Muscle- and bone biopsies
* Quality of life questionnaires
* Testing of muscle funtion
* Metabolic studies of muscle and bone protein turnover using labelling with deuturated water

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60-75 years old, any ethnicity.
* Participants with T- score between < 1.0 and > -2.5 measured by DXA scan within 6 months of the first day of the study.
* Adequate cognitive function to be able to give informed consent.

Exclusion Criteria:

* Osteoporosis and fracture history

  * Participants with osteoporosis (defined by DXA scan < 6 months old: low bone mass, T-score < -2.5 or hip fracture or clinical compression fracture of the spine).
  * History of low energy fractures within last 6 months. Health conditions limiting exercise
  * Health conditions that could limit walking and weightbearing exercise (for instance recent surgery, mobility limitation)
  * Participants with impaired wound healing or history of a chronic open wound Bone metabolism disorders
  * Primary hyperparathyroidism.
  * Known vitamin D deficiency (<25 nM) (re-test after substitution acceptable).
  * Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, severe renal impairment (eGFR < 30) or impaired liver function (baseline phosphatase higher than twice upper limit (105 U/L)), active rheumatic diseases, celiac disease, severe chronic obstructive lung disease (COPD), hypopituitarism, or Cushing's disease.
  * Previous use of bone antiresorptive or bone anabolic drugs within the last 5 years.

Medication use and health conditions

* Use of anabolic steroids in the previous year.
* Use of antiresorptive therapy in the previous year.
* Known medication/supplements affecting bone in the previous year.
* Diabetes type 1 and 2.
* Heart failure similar to NYHA Class IV.
* Treatment with drugs known to affect cytochrome P450 3A due to its role in everolimus metabolism, excluding strong CYP3A4 inhibitors or inducers, while allowing weak and intermediate inhibitors or inducers. Patients on the following drugs will be excluded from the trial: Ketoconazole, Itraconazole, Posaconazole, Voriconazole, Telithromycin, Clarithromycin, Nedazodone, Ritonavir, Atazanavir, Saquinavir, Darunavir, Indinavir, Nelfinavir, Rifampicin, Dexamethasone, Carbamazepine, phenobarbital, Phenytoin, Efavirenz and Nivirapine.
* History of coagulopathy or medical condition requiring long-term anticoagulation.

Blood disorders and other health concerns

* Anemia - Hg < 5,59 mmol/L, Leukopenia - white blood cells (WBC) < 3,5 x 10⁹/L, Neutropenia absolute neutrophil count < 2,0 x 10⁹/L, or Platelet count - platelet count < 125 x 10⁹/L.
* Insufficiently treated dyslipidemia with LDL-c > 4,9 mmol/L and family history of dyslipidemia, Total cholesterol > 9,1 mmol/L, or triglycerides > 9,9 mmol/L.

Immunosuppressive and current cancer Treatment

* Scheduled for immunosuppressant therapy for transplant or scheduled to undergo chemotherapy or any other treatment for malignancy
* Any form of clinically relevant primary or secondary immune dysfunction or deficiency Cardiovascular and heart conditions
* Unstable ischemic heart disease.

Allergies

* Known allergy to rapamycin or rapalogs. Language limitations
* The study will exclude participants with inability to speak and understand Danish and with inability to cooperate.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
P1NP | From baseline to end of treatment at 24 weeks
  Percentage change in circulating levels of bone formation marker N-terminal fragment of procollagen type 1 (P1NP) at 24 weeks as compared with baseline

SECONDARY OUTCOMES:
Bone resorption markers | From baseline to end of treatment 24 weeks
  Change in bone resorption markers (C-terminal telopeptide of type 1 collagen (CTX) at baseline, 4, 12 and 24 weeks.
BMD | From screening to end of treatment 24 weeks
  Lumbar spine (L1-4), and total hip and femoral neck bone mineral density (BMD) measured by dual-energy X-ray absorptiometry (DXA) at screening visit/baseline, and 24 weeks.
Bone mass | From baseline to end of treatment 24 weeks
  Bone mass at the distal radius and tibia measured using high-resolution peripheral quantitative computed tomography (HR-pQCT) at baseline, and 24 weeks.
Bone microarchitecture | From baseline to end of treatment 24 weeks
  Bone microarchitecture at the distal radius and tibia measured using high-resolution peripheral quantitative computed tomography (HR-pQCT) at baseline, and 24 weeks.
Bone geometry | From baseline to end of treatment (24 weeks)
  Bone geometry at the distal radius and tibia measured using high-resolution peripheral quantitative computed tomography (HR-pQCT) at baseline and 24 weeks.
Muscle Cross-Sectional Area | From baseline to end of treatment 24 weeks
  Muscle Cross-Sectional Area (CSA) measured by Magnetic Resonance Imaging (MRI) at baseline, 12, and 24 weeks.
Muscle assessment | From baseline to end of treatment 24 weeks
  Change in muscle strength for the lower extremities, measured using a isokinetic dynamometry at baseline, midway and week 24.
Metabolic health (test 1) | From baseline to end of treatment 24 weeks
  Body weight measured by a digital scale at baseline, 4, 12, and 24 weeks.
Quality of life quiestionaire | From baseline to end of treatment 24 weeks
  Quality of life (QoL)questionnaire SF-12 questionnaire (including mental QoL and physical QoL, and various health and possible side effects) at baseline and 24 weeks
Muscle function (power) | From baseline to end of treatment 24 weeks.
  Muscle function (power) using the 30-second sit-to-stand test (RSS) at baseline, midway and week 24.
Bone formation markers | From baseline to end of study 24 weeks
  P1NP at baseline, 4 and 12 and 24 weeks.
Metabolic health (test 2) | From screening to end of treatment 24 weeks
  Total body fat percentage assessed by dual-energy X-ray absorptiometry (DXA), at screening and 24 weeks.
Metabolic health (test 3) | From baseline to end of treatment 24 weeks
  Lipid parameters (LDL, HDL, Triglycerides, Cholesterol) at baseline, 4, 12, and 24 weeks
Metabolic Health (Test 4) | From screening to end treatment
  Total lean mass assessed by dual-energy X-ray absorptiometry (DXA) screening and baseline, and 24 weeks.
Metabolic health (test 5) | From screening to end of treatment 24 weeks
  Bone mineral density assessed by dual-energy X-ray absorptiometry (DXA) at screening and 24 weeks.

OTHER OUTCOMES:
Biomarkers of biological aging | From baseline to end of treatment 24 weeks
  Measurements of Biomarkers of biological aging in serum: senescence associated secretory phenotype (SASP), which reflect the whole-body burden of senescent cells at baseline and 24 weeks.
Epigenetic clocks | From baseline to end of treatment 24 weeks
  Changes in biological age as determined by "epigenetic clocks" that estimate biological age based on DNA methylation pattern in a selected number of genes. Peripheral blood mononuclear cells (PBMCs) will be isolated from blood at baseline and 24 weeks. DNA will be obtained for DNA methylation evaluation and a fixed part of PBMCs will be used to determine cellular and molecular changes of bone resorbing cells (osteoclast).
Bone changes | At the end of the study 24 weeks
  Two G8 bone biopsies will be obtained at the end of the trial to determine: (a) histomorphometric changes taking place at tissue levels (osteoblastic and osteoclastic activities), (b) global changes in gene expression taking place at tissue level by performing RNA-seq.
  (c) Spatial transcriptomics: measuring changes in gene expression at cellular levels, (d) r nanoindentation and spectroscopies to study bone strength and mineral properties (e) scanned with high resolution CT scanner for determining tissue-levels changes in microarchitecture
Changes in bone stem cell characteristics and the composition of the cells | At the end of the study 24 weeks
  Bone marrow aspirates will be obtained to study changes in bone stem cell (called marrow stromal or mesenchymal stem cells, MSC) characteristics and the composition of the cells within the bone marrow cell population within each treatment arm. Following isolation of MSC, part of the cells will be prepared for single cell RNA-seq to determine changes in cellular composition of bone microenvironment and cellular senescence signature as an estimate of senescent cell burden and the rest will be store for further analysis of the cellular and molecular characteristics e.g. cell proliferation, cell differentiation, changes in metabolic activity. The bone marrow aspirate and bone biopsy samples will be exchanged between the two sites depending on the assays to be performed
Cell size and tissue composition | From baseline to end of treatment 24 weeks
  Muscle biopsies taken at baseline and at 24 weeks: to determine cell size and tissue composition using global proteomic.
Protein turnover in muscle and bone | From baseline to end of treatment 24 weeks
  Muscle biopsies (at baseline and 24 weeks) and bone biopsy (end of study 24 weeks) to determine protein turnover in muscle and bone, respectively from participant agreed to receive deuterium oxide (D2O).

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Kassem, MD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Institute of Sports Medicine, Bispebjerg Hospital, Bispebjerg, Region Sjælland
  - Department of Endocrinology, Odense University Hospital, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No